CLINICAL TRIAL: NCT04758663
Title: The Role of Naps and Overnight Sleep on Cognitive Learning in Preschoolers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Rebecca Spencer, Associate Professor of Psychological and Brain Sciences, University of Massachusetts, Amherst
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-2488
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Within subject comparison of nap/overnight and wake/overnight conditions in habitual and non-habitual nappers
Masking Description: Within-subject; participants/experimenters are aware of conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Declarative memory (Experimental): Napping v. wake effect on declarative memory in habitual and non-habitual nappers.
  Interventions: Behavioral: Nap/wake conditions on memory
- Overnight Physiology (Experimental): Napping v. wake effect on overnight physiology in habitual and non-habitual nappers.
  Interventions: Behavioral: Nap/wake conditions on overnight physiology

INTERVENTIONS:
Behavioral: Nap/wake conditions on memory — Habitual and non-habitual napping children will complete a two conditions-a nap condition where they are encouraged to nap in the afternoon and a wake condition where instead of napping, they spend an equal amount of time awake engaging in quiet activities.
  Arms: Declarative memory
Behavioral: Nap/wake conditions on overnight physiology — Habitual and non-habitual napping children will complete a two conditions-a nap condition where they are encouraged to nap in the afternoon and a wake condition where instead of napping, they spend an equal amount of time awake engaging in quiet activities. On the nights of the nap and wake conditions, physiology will be recorded in habitual and non-habitual nappers.
  Arms: Overnight Physiology

SUMMARY:
The goal of this research is to understand the role of sleep on memory function in early childhood. Specifically, we seek to examine how promoted naps vs. promoted waking in habitual and non-habitual napping children may impact overnight sleep physiology and subsequent memory consolidation.

DETAILED DESCRIPTION:
With time spent awake, sleepiness increases (i.e., sleep pressure; Borbely, 1982). In young adults, naps following sleep deprivation have significantly elevated slow wave activity (SWA; 1-4 Hz) relative to naps following normal overnight sleep (Werth et al., 1996). Similarly in preschool children, overnight sleep following nap deprivation yields significantly greater SWS relative to when a nap was taken earlier in the day (Lassonde et al., 2016). This impact on subsequent sleep physiology suggests that naps may be an extension of overnight sleep. How napping status (i.e., habitual and non-habitual napping) impacts overnight sleep physiology and subsequent memory consolidation is unknown. Thus, this study aims to investigate how napping vs. staying awake in habitual and non-habitual napping children may impact overnight sleep physiology and subsequent memory consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Family lives within 30 miles of UMass Amherst
* Is 33-71 months at the time of enrollment
* Meets the definition of a habitual (5+ naps/week) or non-habitual (<2 naps/week) napper
* Normal or corrected-to-normal vision and hearing
* Access to a computer with an internet connection for online sessions with the research team.

Exclusion Criteria:

* Diagnosis of any sleep disorder (other than mild parasomnia which is routine at this age) past or present
* Current use of psychotropic or sleep-altering medications
* Traveling beyond 1 time zone within 1 month of participation
* Fever or symptoms of respiratory illness at the time of participation
* Diagnosed developmental disability

Ages: 33 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Overnight sleep physiology | 9-11 hours of sleep overnight
  Amount of slow wave activity and other non-REM sleep features in overnight sleep following a day where a nap was involved compared to when there was no nap earlier in the day.

SECONDARY OUTCOMES:
Change in memory accuracy | 2-3 hours/24 hours
  Accuracy on the memory task following the nap compared to before the nap relative to the same memory change measured over an interval spent awake. Further, accuracy on the memory task 24hrs later compared to before the nap/wake interval.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca M Spencer, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No